CLINICAL TRIAL: NCT07311798
Title: Impact of Vascular Resection on Survival and Postoperative Outcomes in Patients With Hilar Cholangiocarcinoma: A Retrospective Study
Status: Not yet recruiting | Type: Observational
Sponsor: Yongjun Chen (Other)
Responsible Party: Sponsor-Investigator, Yongjun Chen, Director, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: BTC-002
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cholangiocarcinoma, Hilar
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vascular Resection Group: Patients with hilar cholangiocarcinoma who underwent curative-intent surgery with concomitant vascular resection, including portal vein and/or hepatic artery resection.
  Interventions: Other: No Intervention: Observational Cohort
- Non-Vascular Resection Group: Patients with hilar cholangiocarcinoma who underwent curative-intent surgery without vascular resection.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — This is an observational study. No intervention is assigned.

SUMMARY:
Hilar cholangiocarcinoma is a highly aggressive malignancy, and surgical resection remains the only potentially curative treatment. Due to the frequent involvement of major vascular structures, vascular resection is increasingly performed to achieve negative surgical margins; however, its impact on survival and postoperative outcomes remains controversial. This retrospective study aims to evaluate the association between vascular resection and clinical outcomes, including survival and postoperative outcomes, in patients with hilar cholangiocarcinoma undergoing curative-intent surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgical treatment at the Department of Hepatobiliary and Pancreatic Surgery of our hospital between January 2010 and December 2024, including those with or without concomitant vascular resection.
* Pathologically confirmed diagnosis of hilar cholangiocarcinoma after surgery.
* Complete clinical and follow-up data available for outcome analysis.

Exclusion Criteria:

* Patients with distant metastasis or who underwent only palliative or exploratory surgery.
* Patients diagnosed preoperatively or intraoperatively with other types of biliary malignancies not located at the hilar region.
* Patients with incomplete medical records or missing key clinical or follow-up data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients who underwent curative-intent surgery for hilar cholangiocarcinoma at the Department of Hepatobiliary and Pancreatic Surgery of our hospital between January 2010 and December 2024. Patients were included regardless of whether vascular resection was performed. All patients had a pathologically confirmed diagnosis of hilar cholangiocarcinoma and sufficient clinical and follow-up data for outcome analysis. Patients with distant metastasis, those who underwent only palliative or exploratory surgery, or those with incomplete medical records or missing key clinical or follow-up information were excluded. According to intraoperative findings, patients were categorized into vascular resection and non-vascular resection cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complications Grade II or Higher (Clavien-Dindo ≥ II) | Within 30 days after surgery
  Postoperative complications within 30 days after surgery will be assessed and classified according to the Clavien-Dindo classification system. Grade II or higher complications are defined as complications requiring pharmacological treatment, blood transfusion, interventional procedures, reoperation, intensive care management, or resulting in death.
Overall Survival (OS) | From surgery to death or last follow-up (up to 5 years)
  Time from the date of curative-intent surgery to death from any cause or last follow-up. Patients who are alive at the last follow-up will be censored. Survival data will be collected from medical records and follow-up visits.

SECONDARY OUTCOMES:
Perioperative Mortality | 30 days after surgery or during hospitalization
  Death occurring within 30 days after surgery or during the index hospitalization, whichever occurs later.
Length of Postoperative Hospital Stay | From the date of surgery to hospital discharge, assessed up to 90 days.
  Number of days from the date of surgery to hospital discharge.
Intraoperative Blood Loss | During surgery
  Estimated blood loss recorded in the operative report, measured in milliliters.
Disease-Free Survival (DFS) | From surgery to tumor recurrence, metastasis, death, or last follow-up (up to 5 years)
  Time from surgery to tumor recurrence, metastasis, death from any cause, or last follow-up, whichever occurs first.